CLINICAL TRIAL: NCT03841162
Title: Fast Assay for Pathogen Identification and Characterization - Prospective Observational Study
Brief Title: Fast Assay for Pathogen Identification and Characterization
Acronym: FAPIC
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other); University of Zagreb (Other); Molzym (Unknown); AIT Austrian Institute of Technology GmbH (Other); BEE Robotics (Unknown); University of Warwick (Other); Claude Bernard University (Other); Axo Science (Unknown)
Responsible Party: Principal Investigator, prof. dr. Inge Gyssens, Principal Investigator, Radboud University Medical Center
Other Study IDs: 18.106/infect18.03
Record Dates: First submitted 2019-02-06; First posted 2019-02-15 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Bacteremia; Sepsis; Septic Shock
Keywords: Blood Cultures
MeSH Terms: conditions — Bacteremia; Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1 EDTA bood sample per blood culture set (2 per patient). 5mL of samples is used for validation of DNA-based diagnostics developed within the FAPIC-project. 4mL of samples is used for HLA-DR typing using flow cytometry. Left-overs are stored as plasma for future research.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected sepsis: Patients for whom blood cultures are drawn at the Emergency Department or the department of Infectious Diseases/Nephrology

SUMMARY:
Sepsis is a life-threatening disease caused by a dysregulated host response to infection. This can lead to organ-dysfunction and septic shock, which is a subset of sepsis where underlying abnormalities increase mortality remarkably. Blood cultures are the gold standard for identifying pathogens in the bloodstream (bacteremia). It is based on cultivation techniques which, theoretically, can detect a single pathogenic cell from a patient sample. However, blood cultures have serious limitations, such as long time to result (3-7 days). This leads to the fact that only a small fraction of the patients obtain a correct diagnosis and in further consequence get the optimal antimicrobial treatment. Patients with sepsis should get antimicrobial treatment within the hour. Thus, physicians start treatment empirically, with broad-spectrum antibiotics. This puts a selective pressure on pathogens and has led to an increased amount of antibiotic resistance. Faster diagnostics are necessary to ensure an immediate and targeted treatment. In the EU-funded FAPIC project, two diagnostic systems that can be used with direct sample material from patients will be developed, avoiding the time-consuming cultivation of pathogens.

In this study, the evaluation of the rapid diagnostics will be performed in patients with sepsis, suspected of bacteremia. To this aim, the performance of the diagnostic systems will be evaluated using blood samples that are collected in parallel with blood cultures. In addition, clinical data of the patients will be collected. In routine care, two blood culture sets (2x2 bottles) per patient are collected. One extra blood samples (EDTA, 9 ml) will be sampled with each blood culture set, totaling 2 samples per patient. In this study, patients presenting at the Emergency Department (ED), and the department of infectious diseases/nephrology will be included. The results will be used to estimate the performance, sensitivity, and specificity of the diagnostic systems compared to blood culture. Furthermore, in order to determine the severity of sepsis and to describe the patient population, clinically relevant parameters and laboratory parameters (ferritin, HLA-DR, serum lactate, SOFA score) will be assessed to determine its association with severity of disease and patient mortality. Evaluation will be done exclusively in the lab, and will not be used directly for the diagnosis or management of patients. Standard care will still be provided.

DETAILED DESCRIPTION:
This study is a follow-up study of the first prospective study performed in 2017 in the same hospital. The ClinicalTrials.gov ID number of the previous study was NCT03025802.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom blood cultures are drawn
* Age ≥ 18

Exclusion Criteria:

* Age < 18
* Patients who are not hospitalized and sent home after ED admission
* Patients from the haematology department
* Duplicate blood cultures from the same bacteraemia episode (blood cultures drawn <7 days after first blood culture)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected sepsis, for whom blood cultures are drawn.
Sampling Method: Probability Sample
Enrollment: 1957 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Confirmed bacteremia based on positive blood cultures (SOFA score) | 7 days
  Differences in SOFA score between patients with positive blood cultures and patients with negative blood cultures.
  SOFA: Sequential Organ Failure Assessment; Range 0-4 (better to worse).
Confirmed bacteremia based on positive blood cultures (Serum Lactate) | 7 days
  Differences in Serum Lactate levels between patients with positive blood cultures and patients with negative blood cultures
Confirmed bacteremia based on positive blood cultures (Ferritin) | 7 days
  Differences in Ferritin levels between patients with positive blood cultures and patients with negative blood cultures
Test performance | 1 year
  Performance characteristics (Clinical sensitivity, specificity and accuracy) of a new rapid diagnostic systems

SECONDARY OUTCOMES:
Length of Stay (SOFA score) | 1 year
  Differences in length of stay between patients with high and with low SOFA score SOFA: Sequential Organ Failure Assessment; Range 0-4 (better to worse).
Length of Stay (Serum Lactate) | 1 year
  Differences in length of stay between patients with high and with low Serum Lactate levels
Length of Stay (Ferritin) | 1 year
  Differences in length of stay between patients with high and with low Ferritin levels
30-day Mortality (Sofa score) | 30 days
  Differences in 30-day mortality between patients with high and with low SOFA score SOFA: Sequential Organ Failure Assessment; Range 0-4 (better to worse).
30-day Mortality (Serum Lactate) | 30 days
  Differences 30-day mortality between patients with high and with low Serum Lactate levels
30-day Mortality (Ferritin) | 30 days
  Differences 30-day mortality between patients with high and with low Ferritin levels

CONTACTS AND LOCATIONS:
Overall Officials: Inge C Gyssens, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Shankar-Hari M, Phillips GS, Levy ML, Seymour CW, Liu VX, Deutschman CS, Angus DC, Rubenfeld GD, Singer M; Sepsis Definitions Task Force. Developing a New Definition and Assessing New Clinical Criteria for Septic Shock: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):775-87. doi: 10.1001/jama.2016.0289. PMID 26903336
- [Background] Faix JD. Biomarkers of sepsis. Crit Rev Clin Lab Sci. 2013 Jan-Feb;50(1):23-36. doi: 10.3109/10408363.2013.764490. PMID 23480440
- [Background] Lvovschi V, Arnaud L, Parizot C, Freund Y, Juillien G, Ghillani-Dalbin P, Bouberima M, Larsen M, Riou B, Gorochov G, Hausfater P. Cytokine profiles in sepsis have limited relevance for stratifying patients in the emergency department: a prospective observational study. PLoS One. 2011;6(12):e28870. doi: 10.1371/journal.pone.0028870. Epub 2011 Dec 29. PMID 22220196
- [Background] Kibe S, Adams K, Barlow G. Diagnostic and prognostic biomarkers of sepsis in critical care. J Antimicrob Chemother. 2011 Apr;66 Suppl 2:ii33-40. doi: 10.1093/jac/dkq523. PMID 21398306
- [Background] Cinel I, Opal SM. Molecular biology of inflammation and sepsis: a primer. Crit Care Med. 2009 Jan;37(1):291-304. doi: 10.1097/CCM.0b013e31819267fb. PMID 19050640
- [Background] Gogos CA, Drosou E, Bassaris HP, Skoutelis A. Pro- versus anti-inflammatory cytokine profile in patients with severe sepsis: a marker for prognosis and future therapeutic options. J Infect Dis. 2000 Jan;181(1):176-80. doi: 10.1086/315214. PMID 10608764
- [Background] Rosario C, Zandman-Goddard G, Meyron-Holtz EG, D'Cruz DP, Shoenfeld Y. The hyperferritinemic syndrome: macrophage activation syndrome, Still's disease, septic shock and catastrophic antiphospholipid syndrome. BMC Med. 2013 Aug 22;11:185. doi: 10.1186/1741-7015-11-185. PMID 23968282
- [Background] Schulert GS, Grom AA. Pathogenesis of macrophage activation syndrome and potential for cytokine- directed therapies. Annu Rev Med. 2015;66:145-59. doi: 10.1146/annurev-med-061813-012806. Epub 2014 Nov 5. PMID 25386930
- [Background] Kell DB, Pretorius E. Serum ferritin is an important inflammatory disease marker, as it is mainly a leakage product from damaged cells. Metallomics. 2014 Apr;6(4):748-73. doi: 10.1039/c3mt00347g. PMID 24549403
- [Background] Carcillo JA, Simon DW, Podd BS. How We Manage Hyperferritinemic Sepsis-Related Multiple Organ Dysfunction Syndrome/Macrophage Activation Syndrome/Secondary Hemophagocytic Lymphohistiocytosis Histiocytosis. Pediatr Crit Care Med. 2015 Jul;16(6):598-600. doi: 10.1097/PCC.0000000000000460. No abstract available. PMID 26154908
- [Background] Bennett TD, Hayward KN, Farris RW, Ringold S, Wallace CA, Brogan TV. Very high serum ferritin levels are associated with increased mortality and critical care in pediatric patients. Pediatr Crit Care Med. 2011 Nov;12(6):e233-6. doi: 10.1097/PCC.0b013e31820abca8. PMID 21263363
- [Background] Kyriazopoulou E, Leventogiannis K, Norrby-Teglund A, Dimopoulos G, Pantazi A, Orfanos SE, Rovina N, Tsangaris I, Gkavogianni T, Botsa E, Chassiou E, Kotanidou A, Kontouli C, Chaloulis P, Velissaris D, Savva A, Cullberg JS, Akinosoglou K, Gogos C, Armaganidis A, Giamarellos-Bourboulis EJ; Hellenic Sepsis Study Group. Macrophage activation-like syndrome: an immunological entity associated with rapid progression to death in sepsis. BMC Med. 2017 Sep 18;15(1):172. doi: 10.1186/s12916-017-0930-5. PMID 28918754
- [Background] Shakoory B, Carcillo JA, Chatham WW, Amdur RL, Zhao H, Dinarello CA, Cron RQ, Opal SM. Interleukin-1 Receptor Blockade Is Associated With Reduced Mortality in Sepsis Patients With Features of Macrophage Activation Syndrome: Reanalysis of a Prior Phase III Trial. Crit Care Med. 2016 Feb;44(2):275-81. doi: 10.1097/CCM.0000000000001402. PMID 26584195
- [Background] Antonakos N, Tsaganos T, Oberle V, Tsangaris I, Lada M, Pistiki A, Machairas N, Souli M, Bauer M, Giamarellos-Bourboulis EJ. Decreased cytokine production by mononuclear cells after severe gram-negative infections: early clinical signs and association with final outcome. Crit Care. 2017 Mar 9;21(1):48. doi: 10.1186/s13054-017-1625-1. PMID 28274246
- [Background] Gainaru G, Papadopoulos A, Tsangaris I, Lada M, Giamarellos-Bourboulis EJ, Pistiki A. Increases in inflammatory and CD14dim/CD16pos/CD45pos patrolling monocytes in sepsis: correlation with final outcome. Crit Care. 2018 Mar 3;22(1):56. doi: 10.1186/s13054-018-1977-1. PMID 29499723
- [Background] Drewry AM, Ablordeppey EA, Murray ET, Beiter ER, Walton AH, Hall MW, Hotchkiss RS. Comparison of monocyte human leukocyte antigen-DR expression and stimulated tumor necrosis factor alpha production as outcome predictors in severe sepsis: a prospective observational study. Crit Care. 2016 Oct 20;20(1):334. doi: 10.1186/s13054-016-1505-0. PMID 27760554
- [Background] Cazalis MA, Friggeri A, Cave L, Demaret J, Barbalat V, Cerrato E, Lepape A, Pachot A, Monneret G, Venet F. Decreased HLA-DR antigen-associated invariant chain (CD74) mRNA expression predicts mortality after septic shock. Crit Care. 2013 Dec 10;17(6):R287. doi: 10.1186/cc13150. PMID 24321376
- [Background] Wang AY, Ma HP, Kao WF, Tsai SH, Chang CK. Red blood cell distribution width is associated with mortality in elderly patients with sepsis. Am J Emerg Med. 2018 Jun;36(6):949-953. doi: 10.1016/j.ajem.2017.10.056. Epub 2017 Nov 10. PMID 29133071
- [Background] Kim CH, Park JT, Kim EJ, Han JH, Han JS, Choi JY, Han SH, Yoo TH, Kim YS, Kang SW, Oh HJ. An increase in red blood cell distribution width from baseline predicts mortality in patients with severe sepsis or septic shock. Crit Care. 2013 Dec 9;17(6):R282. doi: 10.1186/cc13145. PMID 24321201
- [Derived] D'Onofrio V, Heylen D, Pusparum M, Grondman I, Vanwalleghem J, Meersman A, Cartuyvels R, Messiaen P, Joosten LAB, Netea MG, Valkenborg D, Ertaylan G, Gyssens IC. A prospective observational cohort study to identify inflammatory biomarkers for the diagnosis and prognosis of patients with sepsis. J Intensive Care. 2022 Mar 9;10(1):13. doi: 10.1186/s40560-022-00602-x. PMID 35264246
- [Derived] D'Onofrio V, Van Steenkiste E, Meersman A, Waumans L, Cartuyvels R, Van Halem K, Messiaen P, Gyssens IC. Differentiating influenza from COVID-19 in patients presenting with suspected sepsis. Eur J Clin Microbiol Infect Dis. 2021 May;40(5):987-995. doi: 10.1007/s10096-020-04109-x. Epub 2020 Dec 3. PMID 33274416
- See also: FAPIC project website — http://www.fapic.eu